CLINICAL TRIAL: NCT05933850
Title: Culturally Adapted Strong Families Programme to Improve Child Behavior and Family Functioning in Families Living in Gilgit Baltistan, Pakistan
Brief Title: Culturally Adapted Strong Families Programme for Families Living in Gilgit Baltistan, Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: UNODC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PILL-SFP-GB-001
Record Dates: First submitted 2023-05-25; First posted 2023-07-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strong Family Programme Intervention (Experimental): There will be 3 weekly group sessions of the strong family programme with caregivers and children (8-12 families per group).
  Interventions: Behavioral: Strong Families Programme Intervention
- Waitlist control group (Active Comparator): This group will be on the waiting list and receive SF programme training sessions once the study will be completed.
  Interventions: Behavioral: Strong Families Programme Intervention

INTERVENTIONS:
Behavioral: Strong Families Programme Intervention — This is a family skills programme providing an evidence-informed prevention to support caregivers to be better parents and strengthen positive age-specific and age-appropriate family functioning and interactions to help prevent drug use, violence and other negative social consequences in their children.

SUMMARY:
The aim of this exploratory study is to test the Strong Family (SF) programme in improving family functioning when implemented in Gilgit-Baltistan. Participants will be randomized to one of the two study arms 1)- Intervention group in which participants will receive 3 group sessions of SF programme (8-12 families per group) 2)- Control group (control group will be in the waiting list and receive SF training sessions once the study will be completed).

DETAILED DESCRIPTION:
This will be multicentre feasibility randomised controlled trial to test the effectiveness of the SF programme in improving family skills outcomes and caregiver and child mental health, as reported by caregivers when implemented in Gilgit-Baltistan. The study will record families' rates of recruitment and attendance to SF programme, evaluate the completeness of programme delivery, cultural acceptability through qualitative interviews and assess the fidelity of training delivery. A small pilot study with N=10 families (a female caregiver (mother) and one child between the age of 8-15 years from each family) will be conducted before main RCT. The study will be conducted in three districts including; Gilgit, Hunza and Skardu in Gilgit Baltistan, Pakistan. We will interview a subset of participants i.e. up to 5 caregivers from each study site (N=15 caregivers) to explore participants' opinions on the acceptability of the programme and to explore any barriers or facilitators to participation.

ELIGIBILITY:
Inclusion Criteria:

* Female primary caregiver to a child aged between 8-15 years
* Able to speak and understand Urdu language
* Capable to give informed consent

Exclusion Criteria:

* Families that had already taken part in another family skills training programme in the past 6 months or where the caregiver lived separately from the child
* Not the primary caregiver of the child
* Unlikely to be available for the duration of the whole study and outcome assessments (e.g., temporary residence).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Respecting the cultural context, either males or females' caregivers can be engaged at one time in our study setting. As females are most often the primary caregivers in Pakistan, female primary caregivers and their children (of either gender) will be invited to participate in this study.
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability indicators | From baseline to end of intervention at 3 weeks (post randomisation)
  We will record feasibility indicators in terms of families' rates of recruitment and attendance to programme, and programme completeness. To evaluate cultural acceptability of programme by families, interviews with caregivers will be conducted to explore family members' opinions on the acceptability of the programme, any barriers or facilitators to participation.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire | At baseline, week 5 and week 9 of post baseline
  The Strengths and Difficulties Questionnaire is a brief behavioural screening questionnaire and ask about 25 attributes, some positive and others negative. This will be administered to both child and the caregiver.
Parenting and Family Adjustment Scale | At baseline, week 5 and week 9 of post baseline
  This will measures parenting practices and parental adjustment. This scale has been developed to be used in low resource settings.
Child and Youth Resilience Measure | At baseline, week 5 and week 9 of post baseline
  This is a screening tool to explore the resources available that may bolster resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Salman Shahzad, Principal Investigator — Pakistan Institute of Living and Learning

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with other researchers, encompassing essential information such as demographic details, primary and secondary outcome measures, intervention exposure metrics, and process evaluation data. Rigorous measures will be implemented to ensure the complete de-identification of the data and safeguard the anonymity of individual participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After 2 years of trial completion.
Access Criteria: The data could be requested from the corresponding author with a reasonable request.

REFERENCES:
- [Derived] El-Khani A, Asif M, Shahzad S, Bux MS, Maalouf W, Rafiq NUZ, Khoso AB, Chaudhry IB, Van Hout MC, Zadeh Z, Tahir A, Memon R, Chaudhry N, Husain N. Assessing the efficacy of a brief universal family skills programme on child behaviour and family functioning in Gilgit-Baltistan, Pakistan: protocol for a feasibility randomised controlled trial of the Strong Families programme. BMJ Open. 2024 Jul 1;14(6):e081557. doi: 10.1136/bmjopen-2023-081557. PMID 38951006